CLINICAL TRIAL: NCT01166386
Title: An Acute Neurobehavioral Program for Improving Functional Status After TBI
Brief Title: Acute Neurobehavioral Program for Improving Functional Status After TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HD052922-06 (NIH); 1R01HD052922-01A2 (NIH)
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2018-03

CONDITIONS: Traumatic Brain Injury
Keywords: rehabilitation; brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First steps treatment intervention (Experimental): A brief 10-session manualized acute neurobehavioral intervention program will be individually implemented with randomly assigned treatment participants. Session components include injury-related education, enhancement of self-awareness of deficits from the TBI, coping and cognitive skills training, and supported practice. The acronym "FANCI" refers to the name of the program which is First Steps Acute Neurobehavioral and Cognitive Intervention.
  Interventions: Behavioral: FANCI
- standard rehabilitation care (Placebo Comparator): The controls will spend 10 one-half hours with a therapist viewing videos they choose from a menu, some of which have to do with brain injury. The therapist will interact naturally with the controls and occasionally relate the movie or film to brain injury rehabilitation.
  Interventions: Behavioral: FANCI

INTERVENTIONS:
Behavioral: FANCI — comprehensive neurobehavioral sessions with therapist administrating treatment components
  Other Names: First Steps Acute Neurobehavioral and Cognitive Intervention
  Arms: First steps treatment intervention
Behavioral: FANCI — Watching DVDs chosen by participants on various topics.
  Other Names: control condition
  Arms: standard rehabilitation care

SUMMARY:
The specific aims of the proposed study are to 1) evaluate the efficacy of FANCI for improving functional status following treatment using the FIM, 2) examine the impact of FANCI on broader outcome measures of general emotional and behavioral functioning and productive activity in the community as measured post-treatment and at 6-month follow-up, 3) examine contributions of participant injury severity and cognitive status at time of treatment to treatment outcome and treatment response, 4) examine contributions of treatment variables of session topic and mastery, caregiver presence, and concurrent therapies on treatment outcome and treatment response for inpatients with TBI. Primary outcome measure is the (FIM). We will secondarily compare scores on the Disability Rating Scale (DRS), Glasgow Outcome Scale-Extended (GOSE), Rehabilitation Intensity of Therapy Scale (RITS), and Frontal Systems Behavior Scale (FRsBe). Our design is a parallel groups, single-blind, randomized, controlled trial. We will enroll 150 (75 treatment, 75 control) participants. Inclusion Criteria: Mod to Sev TBI based on time to commands, English speaker, Length of stay ≥ 5 days in acute BI rehabilitation Unit, 18 years of age or older, ≥ 79 on GOAT.

DETAILED DESCRIPTION:
More than 1.7 million people a year in the United States begin confronting life with the medical, cognitive, and psychosocial challenges resulting from traumatic brain injury (TBI). A range of cognitive impairments commonly observed following injury increase caregiver burden as well as per-person lifetime costs for care and support of survivors of TBI, estimated at $600,000 to $1,875,000. Our long-term goal is to lessen these burdens through improving the functional status of patients with TBI by providing an evidence-based, comprehensive, brief, acute-care intervention, First Steps Acute Neurobehavioral and Cognitive Intervention (FANCI). The 10-sesson, manualized FANCI Program will be tested in a controlled, randomized study. Therapeutic components of the FANCI include didactics, cognitive remediation, demonstration, guided self-reflection, rehearsal, and supported practice of skills and strategies. Specific hypotheses are that 1) FANCI will result in more improvement in functional status compared to standard interdisciplinary rehabilitation treatment and 2) FANCI will result in more improvement on measures of neurobehavioral functioning compared to standard rehabilitation care for patients with moderate to severe TBI. We base these hypotheses on the observations that 1) providing information about symptoms, treatment, and coping results in reduced symptom intensity and duration for patients with TBI, and 2) inpatient participants in recent FANCI pilot studies learned >80% of the FANCI Program curriculum, and 3) the most recent pilot study participants had significantly better functional outcomes at discharge than matched controls. The specific aims of the proposed study are to 1) evaluate the efficacy of FANCI for improving functional status following treatment using the FIM, 2) examine the impact of FANCI on broader outcome measures of general emotional and behavioral functioning and productive activity in the community as measured post-treatment and at 6-month follow-up, 3) examine contributions of participant injury severity and cognitive status at time of treatment to treatment outcome and treatment response, 4) examine contributions of treatment variables of session topic and mastery, caregiver presence, and concurrent therapies on treatment outcome and treatment response for inpatients with TBI. Primary outcome measure is the (FIM). We will secondarily compare scores on the Disability Rating Scale (DRS), Glasgow Outcome Scale-Extended (GOSE), Rehabilitation Intensity of Therapy Scale (RITS), and Frontal Systems Behavior Scale (FRsBe). Our design is a parallel groups, single-blind, randomized, controlled trial. We will enroll 150 (75 treatment, 75 control) participants. Inclusion Criteria: Mod to Sev TBI based on time to commands, English speaker, Length of stay ≥ 5 days in acute BI rehabilitation Unit, 18 years of age or older, ≥ 79 on GOAT.

ELIGIBILITY:
Inclusion Criteria: at least 18 years old, English speaking, traumatic brain injury inpatient, out of post traumatic amnesia, not psychotic -

Exclusion Criteria: Prisoner, psychotic, not medically stable

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet P Niemeier, Ph.D., Principal Investigator — Carolinas Rehabilitation, Carolinas Healthcare System
Locations (1):
- Carolinas Rehabilitation, Carolinas Medical Center, Department of Physical Medicine and Rehabilitation, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | First Steps Treatment Intervention | Standard Rehabilitation Care
Started | 82 | 83
Completed | 79 | 78
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Steps Treatment Intervention | Standard Rehabilitation Care | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.62 (16.75) | 42.21 (18.95) | 41.07 (18.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 59 | 58 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 79 | 79 | 158
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 21 | 45
  White | 52 | 57 | 109
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 82 | 83 | 165

OUTCOME MEASURES:

1. Primary Outcome: Functional Independence Measure Scores
Description: Minimum score = 18 Maximum possible with FIM = 126 directionality is toward the level of independence, lower numbers signify greater dependence on help from another person to complete the task or activity
Time Frame: Pre, at end of treatment up to one week, six-month follow up
Population: Several persons terminated the intervention project, some files did not get transferred from one of the PIs institutions to another when she changed jobs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | First Steps Treatment Intervention | Standard Rehabilitation Care
Number analyzed (Participants) | 73 | 70
units on a scale
  baseline | 88.11 (10.26) | 89.79 (12.29)
  at end of treatment up to one week: number analyzed (Participants) | 53 | 48
  at end of treatment up to one week | 120.57 (7.32) | 119.67 (8.03)
  six month follow-up | 48.98 (16.65) | 50.93 (14.86)

2. Secondary Outcome: Neurobehavioral Rating Scale
Description: The Neurobehavioral Rating Scale (NRS) is a provider or family rating scale for describing cognition, emotional, behavioral characteristics of a patient with brain injury. Twenty-seven items assess symptoms such as Fatigueability, Depressive Mood, and Tension with 7-point rating scale including "not present," "Very mild," "Mild," "Moderate," "Mod-Severe," "Severe," and "Extremely Severe" to describe the person being rated. Higher scores indicate worse severity of symptoms and lower score indicate an absence of the symptom or very mild symptomatology. The minimum total score is 27 and the maximum total score is 189. For each individual scale within the measures, the minimum score is 1 and the maximum score is 7.
Time Frame: Pre, post, six month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | First Steps Treatment Intervention | Standard Rehabilitation Care
Number analyzed (Participants) | 73 | 69
units on a scale
  baseline | 56.23 (12.83) | 58.70 (13.60)
  post-treatment | 48.4857 (9.94003) | 50.2985 (10.51264)
  follow-up | 48.9778 (16.64808) | 50.9318 (14.85495)

ADVERSE EVENTS:
Arm/Group | First Steps Treatment Intervention | Standard Rehabilitation Care
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/83
Other Adverse Events (participants affected / at risk) | 0/82 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First Steps Treatment Intervention (N=82) | Standard Rehabilitation Care (N=83)
stroke (Nervous system disorders) | 1 | 0 — Patient passed away at home, three weeks after hospital discharge. Patient's onset was not related to study intervention.

LIMITATIONS AND CAVEATS:
3 treatment subjects were discharged prior to completion of the treatment intervention. 5 controls were discharged prior to completion of the treatment intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes